CLINICAL TRIAL: NCT03099642
Title: Emergency Physician Performed Ultrasound-Assisted Lumbar Puncture in a Pediatric Population: A Randomized Controlled Trial
Brief Title: Ultrasound-Assisted Lumbar Puncture in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, MSc, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UALP
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Fever
Keywords: lumbar puncture; Point of care ultrasound; children
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound assisted lumbar puncture (Experimental): The intervention of interest will be the ultrasound-assisted lumbar puncture (UALP). To do this, the treating physician will perform a bedside ultrasound of the spine to identify and mark the level of the conus medullaris and preferred puncture site prior to LP
  Interventions: Radiation: ultrasound-assisted lumbar puncture
- Standard lumbar puncture (No Intervention): The control group will have a standard landmark-based lumbar puncture

INTERVENTIONS:
Radiation: ultrasound-assisted lumbar puncture — The ultrasound probe type will be selected by the treating pediatric emergency physician who has been trained according to standards outlined below. They will first identify the conus medullaris and make a horizontal marking with a sterile pen on the patient's back. Using a transverse view, they will then identify the midline of the patient's spine (using adjacent spinous processes) and will make 2 vertical skin markings on either side of the probe. Next, they will orient the probe in a longitudinal view to identify the desired vertebral interspace and will make 2 horizontal skin markings on either side of the probe at this level. Finally the 4 lines will be joined together at an intersection point, which will be the predetermined site for puncture attempt.
  Arms: Ultrasound assisted lumbar puncture

SUMMARY:
The aim of this study is to determine if emergency physician performed ultrasound-assisted lumbar puncture improves first-time success rates in a pediatric population. This will be done by comparison with current landmark-based approach to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient less than 19 years of age
* Requiring a lumbar puncture as part of their work-up, as determined by the treating pediatric emergency physician.

Exclusion Criteria:

* • Patients with known spine or spinal cord abnormalities

  * Patients with ventricular shunts
  * Patients deemed too unstable to have procedure performed
  * Patients at risk for significant bleeding (coagulopathy, thrombocytopenia, etc)
  * Parents unable to give consent or patients unable to assent for an acute reason

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 166 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
First-tie success | 15 minutes
  First-time lumbar puncture success rate is defined by the presence of at least 0.5 mL of cerebrospinal fluid with red blood cell count < 1,000/mm3.

SECONDARY OUTCOMES:
Total lumbar puncture success rate | 15 minutes
  defined by the presence of at least 0.5 mL of cerebrospinal fluid with red blood cell count < 1,000/mm3 in any number of attempt
Change in performer | 15 minutes
  If the lumbar puncture was attempted by a second person following the first attempts
Time of procedure | 30 minutes
  Time to perform the lumbar puncture
Complication | 30 minutes
  Occurence of any complication

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Gravel, MD, MSc, Principal Investigator — Sainte-Justine Hospital
Locations (1):
- Sainte-Justine Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No